CLINICAL TRIAL: NCT03517176
Title: A Phase 1 Clinical Trial of CEND-1 in Combination With Nabpaclitaxel and Gemcitabine in Metastatic Exocrine Pancreatic Cancer
Brief Title: CEND-1 in Combination With Nabpaclitaxel and Gemcitabine in Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CEND1-001; U1111-1213-3234 (Other: The Universal Trial Number (UTN))
Record Dates: First submitted 2018-03-15; First posted 2018-05-07 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Dose Escalation) (Experimental): Safety of ascending dose levels of CEND-1 in combination with gemcitabine and nab-paclitaxel will be evaluated. Patients will receive an IV bolus of CEND-1 on Day 1 of the 1-week run-in period. This is followed by one treatment cycle (28 days) with the CEND-1 / nab-paclitaxel (125mg/m^2) / gemcitabine (1000mg/m^2) combination given on Days 1, 8, 15.
  Interventions: Drug: CEND-1; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Part B (Expansion) (Experimental): Safety and early efficacy of CEND-1 in combination with nab-paclitaxel (125mg/m^2) and gemcitabine (1000mg/m^2) will be evaluated (dosing on Days 1, 8, 15 of the 28-day treatment cycle). Treatment cycles will be repeated every 4 weeks based on toxicity and response. Treatment may continue as long as there is perceived benefit or until disease progression.
  Interventions: Drug: CEND-1; Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: CEND-1 — CEND-1 will be provided as concentrate for solution to be administered via IV injection.
  Other Names: LSTA1; certepetide
Drug: Nab-paclitaxel — Nab-paclitaxel will be provided as solution to be administered via IV infusion.
  Other Names: Abraxane
Drug: Gemcitabine — Gemcitabine will be provided as solution to be administered via IV infusion.
  Other Names: Gemzar

SUMMARY:
CEND-1, Gemicitabine and Nab-Paclitaxel for Pancreatic Ductal Adenocarcinoma

DETAILED DESCRIPTION:
This is an open-label, multicenter, dose-escalation, safety, pharmacodynamic, pharmacokinetic study of CEND-1 in combination with nabpaclitaxel and gemcitabine administered weekly for three weeks followed by one week off over 28 days.

This protocol is designed to evaluate the safety, tolerability, and biologic activity of CEND-1 in patients with metastatic pancreatic ductal adenocarcinoma (PDAC) who are undergoing combination therapy with nabpaclitaxel and gemcitabine. CEND-1 is a tumor-penetrating peptide (scientifically also known as iRGD) that activates a drug transport mechanism specifically in tumors.

Study involves an initial dose escalation phase with four different CEND-1 dose levels, first as a monotherapy (during 1-week run-in), followed by combination therapy with nabpaclitaxel and gemcitabine (one 28-day treatment cycle). A subsequent expansion phase with approximately 28 subjects will assess the safety, tolerability and preliminary efficacy of the combination treatment using two different CEND-1 dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic pancreatic ductal carcinoma
* One or more metastatic lesions measurable on MRI, PET/CT, or dedicated CT scan according to RECIST v1.1.
* Eligible for treatment with nabpaclitaxel and gemcitabine
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 3 months
* Adequate archival tissue from prior biopsy for biomarker evaluation or willingness to undergo biopsy before treatment starts
* The patient is capable of understanding and complying with the protocol and the subject or, when applicable, the subject's legally acceptable representative has signed the informed consent
* A negative serum pregnancy test (if a premenopausal female patient)
* Acceptable liver function: Bilirubin ≥ 1.5 times upper limit of normal; AST (SGOT) < 10 times upper limit of normal, ALT (SGPT) and Alkaline phosphatase 2.5 times upper limit of normal (if liver metastases are present, then ≤ 5 x ULN is allowed).
* Acceptable renal function: Serum creatinine within normal limits; calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal by the Cockroft-Gault equation.
* Acceptable hematologic status: Granulocyte ≥ 1500 cells/mm3; Platelet count ≥ 100,000 plt/mm3; Hemoglobin ≥ 9 g/dL.
* Urinalysis: No clinically significant abnormalities.
* Acceptable coagulation status: PT within normal limits; PTT within normal limits.
* For men and women of child-producing potential, the use of effective contraceptive methods during the study.

Exclusion Criteria:

* Prior chemotherapy or any other investigational agents for the treatment of pancreatic cancer.
* Concurrent use of any other anti-cancer therapy, including chemotherapy, targeted therapy, immunotherapy, or biological agents.
* Participants with known brain metastases.
* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Pregnant or nursing women. Women of child-bearing potential and men must agree to use adequate contraception.
* Unwillingness or inability to comply with procedures required in this protocol.
* Known infection with HIV, hepatitis B, or hepatitis C.
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions per physician judgement) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Safe doses of CEND-1 when given alone or in combination with nabpaclitaxel and gemcitabine | Escalation Phase: From Day 1 of the run-in until Day 28 of Cycle 1 (cycle length=28 days)
  Safety and toxicity profile of treatment regimen as measured by grade and frequency of adverse events, graded and documented according to the NCI CTCAE, version 5.0 guidelines
Optimal Biological Dose (OBD) of CEND-1 when given in combination | Expansion Phase: from baseline until treatment discontinuation and approximately 30 days after last dose (cycle length=28 days)
  OBD will be determined by evaluating biomarkers (such as the tumor marker CA19-9 Response Rate), the ECOG Performance Status and the Disease Control Rate

SECONDARY OUTCOMES:
Pharmacokinetics of CEND-1 when given alone or in combination with nabpaclitaxel and gemcitabine | Escalation phase: Predose, 3 minutes, 15 min, 30 min, 1 h, 4 h, 8 h postdose on Day 1 of the run-in and Day 1 of Cycle 1
  Area Under the Concentration-Time Curve of CEND-1 Following Intravenous (IV) Administration
Disease Control Rate (Complete Remission (CR) + Partial Remission (PR) + Stable Disease (SD)) associated with the administration of CEND-1 in combination with nabpaclitaxel and gemcitabine | Expansion Phase: from baseline until treatment discontinuation and approximately 30 days after last dose (cycle length=28 days)
Preliminary evidence of anti-tumor activity of CEND-1 when given in combination with nabpaclitaxel bound and gemcitabine by objective radiographic assessment according to RECIST 1.1 | Expansion Phase: from baseline until treatment discontinuation and approximately 30 days after last dose (cycle length=28 days)

OTHER OUTCOMES:
Immunohistochemical assessment of tumor biopsies for the expression of Neuropilin-1 in order to study if the response to CEND-1 therapy can be predicted based on the Neuropilin-1 expression level | Screening Phase (Day -14 until Day -1)
  Analysis of paraffin-embedded tumor tissues (also potentially in liquid-nitrogen frozen tissue, if available) will be performed to characterize Neuropilin-1 expression by immunohistochemistry (IHC) and potentially other analysis techniques.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Queen Elizabeth Hospital, Woodville South, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - St John of God Hospital, Subiaco, Western Australia

REFERENCES:
- [Derived] Dean A, Gill S, McGregor M, Broadbridge V, Jarvelainen HA, Price T. Dual alphaV-integrin and neuropilin-1 targeting peptide CEND-1 plus nab-paclitaxel and gemcitabine for the treatment of metastatic pancreatic ductal adenocarcinoma: a first-in-human, open-label, multicentre, phase 1 study. Lancet Gastroenterol Hepatol. 2022 Oct;7(10):943-951. doi: 10.1016/S2468-1253(22)00167-4. Epub 2022 Jul 6. PMID 35803294